CLINICAL TRIAL: NCT06507592
Title: In Vivo Evaluation of the Differences in Oxidative-reductive Processes in Saliva During Treatment With Conventional Brackets and Clear Aligners
Brief Title: Oxidative-reductive Processes and the Degree of Inflammation in Saliva With Conventional Brackets and Clear Aligners
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Vincenzo Grassia, Associate Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: N. Prot. 0637
Record Dates: First submitted 2024-06-03; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Inflammation; Oxidative Stress; TNF-α
Keywords: clear aligners; fixed appliances; oxidative stress; inflammation; orthodontic treatment
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed Appliances (FA) (Other): 13 patients with fixed appliances, between 10 and 18 years of age, with good oral hygiene and without gingival inflammation, has been recruited
  Interventions: Diagnostic Test: Saliva samples collection
- Clear Aligners (CA) (Other): 13 patients with clear aligners, between 10 and 18 years of age, with good oral hygiene and without gingival inflammation, has been recruited
  Interventions: Diagnostic Test: Saliva samples collection

INTERVENTIONS:
Diagnostic Test: Saliva samples collection — The first sample of saliva was be taken before the start of the treatment and considered as the control sample (T0); the second sample was be taken one month after the start of the treatment (T1) and the third one after three months (T2).

SUMMARY:
The purpose of this prospective observational study is to evaluate the differences in oxidative-reductive processes and the degree of inflammation in saliva during treatment with conventional brackets and clear aligners. The evaluation will be performed by determining the salivary values of Total oxidant status (TOS), total antioxidant status (TAS) and 8-hidroxy-2'-deoxyguanosine (8OHdG).

DETAILED DESCRIPTION:
The differences between production of free radicals and the antioxidant capacity of a system is called oxidative stress, this leads oxidative damages to macromolecules, including lipids and proteins.

Oxidative stress occurs in the tissues when the normal balance between ROS production (extracellular Reactive Oxygen Species) and the antioxidant defense shifts in favor of the first; this situation can result from an excess of ROS and/or the reduction of antioxidants. Some ROS types (e.g. superoxide and hydroxyl radicals, hydrogen peroxide, hypochlorous acid) are capable to directly damage proteins, carbohydrates, DNA and lipids; furthermore, ROS production and an altered redox state of tissues can modulate the expression of a variety of immune and inflammatory molecules through redox sensitive transcription factors (eg NF-kB, AP-1), causing thus indirect tissue damage such as inflammation.

Antioxidants agents are found in all biological species to protect against the potential harmful effects of processes or reactions that cause excessive oxidation. Therefore, biological antioxidants represent an important part of our diet and, together with intracellular antioxidants and antioxidant enzyme systems, may prevent various diseases. Antioxidant defense systems are very complex and for this reason it is essential to evaluate the quantity and / or activity of the different systems when evaluating their in vivo state.

Studies on the antioxidant defense systems present in saliva and their relationship with oral diseases are still few. Despite markers of oxidative stress have been found in saliva in presence of systemic and oral diseases, including inflammatory diseases such as gingivitis, periodontitis, caries and oral cancer.4, 15 During an orthodontic treatment, which often lasts for years, some components of the used orthodontic appliance can be released into the oral environment and saliva. The release of these components and their diffusion can cause various adverse effects in the body, such as allergic reactions, systemic toxicity, cytotoxicity, mutagenicity and carcinogenicity. Although there has been satisfactory development of orthodontic materials, the biocompatibility of these materials is usually not well known. The evaluation of these characteristics of orthodontic materials is as important aspect as their physiological or mechanical properties. However, the studies on these characteristics are limited, and they are mostly related to the cytotoxic effects of orthodontic adhesives. The total state of the oxidant (TOS) and the antioxidant (TAS) reflects the oxidative state and provides information on the body's antioxidant capacity. Oxidative damage to DNA can be detected by chemical, physical and enzymatic methods. 8-hydroxyoxiguanosin (8-OHdG) is an oxidized nucleoside which is excreted in body fluids for DNA repair. Several studies have shown that 8-OHdG in body fluids can act as a biomarker of oxidative stress and 8-OHdG is commonly used as a marker to evaluate oxidative DNA damage in disorders including chronic inflammatory diseases. Previous studies have in fact indicated a possible relationship between the salivary levels of 8-OHdG and the diseased periodontium. However, the levels of TOS, TAS and 8-OHdG in patients undergoing therapy with conventional brackets and with clear aligners has not yet been studied.

ELIGIBILITY:
Inclusion Criteria:

* age between 10 and 18 years
* patients with no orthodontic devices in the mouth
* patients requiring orthodontic treatment
* patients who have good oral hygiene
* patients without gingival inflammation

Exclusion Criteria:

* patients with systemic diseases or infections
* patients with previous orthodontic treatments
* patients on drugs or assuming alcohol
* smoking patients
* patients with enamel decalcification or fillings

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-12-21 (Estimated)

PRIMARY OUTCOMES:
Oxidative-reduction and inflammation | One year
  The Total Antioxidant Status (TAS) in saliva samples was measured using a N 2 615700-1KIT Total Antioxidant Status Assay Kit, a colorimetric assay for antioxidant levels in serum or plasma. The Total Oxidant Status (TOS) was measured with a CS0790-1KT Antioxidant Assay Kit, which includes all necessary reagents to measure total antioxidant capacity in plasma, serum, urine, saliva, cells, and tissue lysates. It also measures the radical cation (ABTS+) scavenging capacity. The 8-Hydroxy-2'-deoxyguanosine (8-OHdG) and Tumor Necrosis Factor-α (TNF-α) levels were determined using an E-EL-H0109 HUMAN TNF-ALPHA ELISA KIT, which detects protein levels quantitatively in serum, plasma, or cell lysate supernatants.

SECONDARY OUTCOMES:
Potential risk factors | Two years
  Using plastic-based or metallic materials for orthodontic devices can increase saliva's oxidative and inflammatory status, potentially correlating with conditions like gingivitis, dental caries, periodontitis, or minor lesions such as aphthous ulcers. Oxidative stress impairs the ability to counteract further pathological events. Free radicals or reactive oxygen species (ROS) are typically generated during biochemical redox reactions as part of normal cell metabolism (for protection against infectious agents) and in response to environmental factors like UV radiation, cigarette smoke, pollutants, and gamma radiation. Once formed, ROS can attack cellular components in the mouth, damaging lipids, proteins, and DNA in oral tissues. This damage can initiate or exacerbate oral diseases, including gingivitis, dental caries, periodontitis, and other inflammatory conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Grassia, DDs, PhD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Multidisciplinary Department of Medical-Surgical and Dental Specialties, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
anyone can contact the PI by mail and ask two share the IPD. All data will be stored in a cloud available by University of Campania. The PI will share a link to accede to the files.
Supporting Information: Study Protocol, CSR
Time Frame: The data will be available after paper publication for at least 2 years
Access Criteria: Person involved in research and affiliated in recognized Institution

REFERENCES:
- [Background] Schipper RG, Silletti E, Vingerhoeds MH. Saliva as research material: biochemical, physicochemical and practical aspects. Arch Oral Biol. 2007 Dec;52(12):1114-35. doi: 10.1016/j.archoralbio.2007.06.009. Epub 2007 Aug 10. PMID 17692813
- [Background] Kovac V, Poljsak B, Perinetti G, Primozic J. Systemic Level of Oxidative Stress during Orthodontic Treatment with Fixed Appliances. Biomed Res Int. 2019 May 23;2019:5063565. doi: 10.1155/2019/5063565. eCollection 2019. PMID 31240214
- [Background] Angelieri F, Carlin V, Martins RA, Ribeiro DA. Biomonitoring of mutagenicity and cytotoxicity in patients undergoing fixed orthodontic therapy. Am J Orthod Dentofacial Orthop. 2011 Apr;139(4 Suppl):e399-404. doi: 10.1016/j.ajodo.2009.06.029. PMID 21435548
- [Background] Guler C, Toy E, Ozturk F, Gunes D, Karabulut AB, Otlu O. Evaluation of salivary total oxidant-antioxidant status and DNA damage of children undergoing fixed orthodontic therapy. Angle Orthod. 2015 Mar;85(2):239-44. doi: 10.2319/110113-798.1. Epub 2014 Jun 20. PMID 24949910
- [Background] Krifka S, Hiller KA, Spagnuolo G, Jewett A, Schmalz G, Schweikl H. The influence of glutathione on redox regulation by antioxidant proteins and apoptosis in macrophages exposed to 2-hydroxyethyl methacrylate (HEMA). Biomaterials. 2012 Jul;33(21):5177-86. doi: 10.1016/j.biomaterials.2012.04.013. Epub 2012 Apr 24. PMID 22534037
- [Background] Ambati M, Rani KR, Reddy PV, Suryaprasanna J, Dasari R, Gireddy H. Evaluation of oxidative stress in chronic periodontitis patients following systemic antioxidant supplementation: A clinical and biochemical study. J Nat Sci Biol Med. 2017 Jan-Jun;8(1):99-103. doi: 10.4103/0976-9668.198366. PMID 28250683
- [Background] Ichiishi E, Li XK, Iorio EL. Oxidative Stress and Diseases: Clinical Trials and Approaches. Oxid Med Cell Longev. 2016;2016:3458276. doi: 10.1155/2016/3458276. Epub 2016 Oct 19. No abstract available. PMID 27833701
- [Background] Chiou CC, Chang PY, Chan EC, Wu TL, Tsao KC, Wu JT. Urinary 8-hydroxydeoxyguanosine and its analogs as DNA marker of oxidative stress: development of an ELISA and measurement in both bladder and prostate cancers. Clin Chim Acta. 2003 Aug;334(1-2):87-94. doi: 10.1016/s0009-8981(03)00191-8. PMID 12867278
- [Background] Evans MD, Dizdaroglu M, Cooke MS. Oxidative DNA damage and disease: induction, repair and significance. Mutat Res. 2004 Sep;567(1):1-61. doi: 10.1016/j.mrrev.2003.11.001. PMID 15341901
- [Background] undefined
- [Background] Kaplan MD, Baum BJ. The functions of saliva. Dysphagia. 1993;8(3):225-9. doi: 10.1007/BF01354542. PMID 8359042
- [Background] Cuevas-Cordoba B, Santiago-Garcia J. Saliva: a fluid of study for OMICS. OMICS. 2014 Feb;18(2):87-97. doi: 10.1089/omi.2013.0064. Epub 2014 Jan 3. PMID 24404837
- [Background] Humphrey SP, Williamson RT. A review of saliva: normal composition, flow, and function. J Prosthet Dent. 2001 Feb;85(2):162-9. doi: 10.1067/mpr.2001.113778. PMID 11208206
- [Background] Takane M, Sugano N, Iwasaki H, Iwano Y, Shimizu N, Ito K. New biomarker evidence of oxidative DNA damage in whole saliva from clinically healthy and periodontally diseased individuals. J Periodontol. 2002 May;73(5):551-4. doi: 10.1902/jop.2002.73.5.551. PMID 12027259
- [Background] Sezer U, Cicek Y, Canakci CF. Increased salivary levels of 8-hydroxydeoxyguanosine may be a marker for disease activity for periodontitis. Dis Markers. 2012;32(3):165-72. doi: 10.3233/DMA-2011-0876. PMID 22377732
- [Background] Kumar D, Pandey RK, Agrawal D, Agrawal D. An estimation and evaluation of total antioxidant capacity of saliva in children with severe early childhood caries. Int J Paediatr Dent. 2011 Nov;21(6):459-64. doi: 10.1111/j.1365-263X.2011.01154.x. Epub 2011 Jul 1. PMID 21718374
- [Background] Beyersmann D, Hartwig A. Carcinogenic metal compounds: recent insight into molecular and cellular mechanisms. Arch Toxicol. 2008 Aug;82(8):493-512. doi: 10.1007/s00204-008-0313-y. Epub 2008 May 22. PMID 18496671
- [Background] Canakci CF, Canakci V, Tatar A, Eltas A, Sezer U, Cicek Y, Oztas S. Increased salivary level of 8-hydroxydeoxyguanosine is a marker of premature oxidative mitochondrial DNA damage in gingival tissue of patients with periodontitis. Arch Immunol Ther Exp (Warsz). 2009 May-Jun;57(3):205-11. doi: 10.1007/s00005-009-0026-9. Epub 2009 May 29. PMID 19479201
- [Background] Manuelli M, Marcolina M, Nardi N, Bertossi D, De Santis D, Ricciardi G, Luciano U, Nocini R, Mainardi A, Lissoni A, Abati S, Lucchese A. Oral mucosal complications in orthodontic treatment. Minerva Stomatol. 2019 Apr;68(2):84-88. doi: 10.23736/S0026-4970.18.04127-4. PMID 30854838